CLINICAL TRIAL: NCT05949723
Title: Development of Artificial Intelligence Golf Training Simulator: Integration of Inertial Sensing Device and Musculoskeletal Simulation Model for Movement Feedback System
Brief Title: Development of Artificial Intelligence Golf Training Simulator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202206046RIPA
Record Dates: First submitted 2022-09-26; First posted 2023-07-18 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2023-06

CONDITIONS: Musculoskeletal Model

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Golf simulator device training (Experimental)
  Interventions: Device: Golf simulator device

INTERVENTIONS:
Device: Golf simulator device — The golf simulator can accurately predict the flight trajectory and landing point of the ball using high-speed moving object measurement technology, giving the user the impression that they are playing on a real golf course.

SUMMARY:
The golf simulator can accurately predict the flight trajectory and landing point of the ball using high-speed moving object measurement technology, giving the user the impression that they are playing on a real golf course.

DETAILED DESCRIPTION:
The golf simulator can accurately predict the flight trajectory and landing point of the ball using high-speed moving object measurement technology, giving the user the impression that they are playing on a real golf course. This project will integrate golf simulators, swing analysis, and musculoskeletal simulation systems; digitize human movements; calculate biomechanical parameters; and assist beginners in swing learning or professional golfer training.

ELIGIBILITY:
Inclusion Criteria:

* Healthy golf players and more than 3 years of golf experience
* Age between 20~60 years old

Exclusion Criteria:

* Musculoskeletal disease within 6 months

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-04-14 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Kinematics data_range of motion | 6 months
  A motion capture system is used to measure the joint kinematics. This data is used to calculate the range of motion of each joint of the body (unit: degree) during the golf swing motion.
Kinematics data_displacement of center of mass | 6 months
  A motion capture system is used to measure the joint kinematics. This data is used to calculate the displacement of the center of mass in space (unit: cm) during the golf swing motion.
Kinetic data_mean velocity | 6 months
  The participants stand on the force platform. The data from the force platform is used to calculate the mean velocity of center of pressure (unit: cm/s): total excursion/total time during the golf swing motion.
Kinetic data_mean distance | 6 months
  The participants stand on the force platform. The data from the force platform is used to calculate the mean distance of center of pressure (unit: cm): how far the sway from the center during the golf swing motion.
Kinetic data_mean frequency | 6 months
  The participants stand on the force platform. The data from the force platform is used to calculate the mean frequency of center of pressure (unit: Hz): how vibrating of the sway during the golf swing motion.
Kinetic data_95% confidence ellipse area | 6 months
  The participants stand on the force platform. The data from the force platform is used to calculate 95% confidence ellipse area of center of pressure (unit: cm^2): how big of the sway during the golf swing motion.
Kinematics data by inertial measurement units_linear acceleration | 6 months
  Inertial measurement units are placed on each body segment and are used to calculate the linear acceleration (m/s²) of each body part during the golf swing motion.
Kinematics data by inertial measurement units_angular velocity | 6 months
  Inertial measurement units are placed on each body segment and are used to calculate the angular velocity (rad/s) of each body part during the golf swing motion.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No